CLINICAL TRIAL: NCT04125537
Title: Pathways Project Collaborative Phase II: Implementation of Kidney Supportive Care in Practice
Brief Title: Pathways Project: Kidney Supportive Care
Status: Completed | Type: Observational
Sponsor: George Washington University (Other)
Collaborators: West Virginia University Research Corporation (Unknown); Gordon and Betty Moore Foundation (Other); Coalition for Supportive Care of Kidney Patients (Unknown); Stanford University (Other)
Responsible Party: Principal Investigator, Dale Lupu, PI, George Washington University
Other Study IDs: 180679
Record Dates: First submitted 2019-08-05; First posted 2019-10-14 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Kidney Diseases; Chronic Kidney Diseases; End Stage Renal Disease; End Stage Renal Disease on Dialysis; Chronic Kidney Disease Requiring Chronic Dialysis
Keywords: Shared-Decision Making; Supportive Kidney Care; Goals of Care Conversations; Palliative Care; Palliative Medicine; Advanced Care Planning; Medical Management without Dialysis; Palliative Dialysis; Conservative Kidney Management
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dialysis Centers - Seriously Ill patients - pre-implementation cohort: Dialysis center patients who screened positive as seriously ill in month 1 of the collaborative activities (the preimplementation period).
- Dialysis Centers - Seriously Ill patients - post-intervention cohort: Dialysis Center patients who screened positive as seriously ill in month 15 of the intervention (the post-implementation period).
  Interventions: Behavioral: IHI Breakthrough Collaborative Model

INTERVENTIONS:
Behavioral: IHI Breakthrough Collaborative Model — Staff teams at participating dialysis centers take part in a quality improvement/collaborative learning model that was initially planned to include three in-person learning sessions, and three activity sessions during which staff teams at each site use quality improvement processes to implement kidney supportive care best practices from the change package. Technical assistance, education, and quality improvement coaching are provided to the site staff teams throughout the project. Patients at the sites then receive care that has been improved via this staff education and quality improvement activities.
  Groups: Dialysis Centers - Seriously Ill patients - post-intervention cohort

SUMMARY:
The Pathways Collaborative is the first attempt to implement supportive (palliative) kidney care at multiple sites in the United States. While supportive kidney care is growing in other countries, notably Canada, Australia, and Great Britain, it is not yet known how to integrate it into the unique nephrology environment in the United States. In Phase 1 of Pathways (completed), we developed an evidence-based change packet of 14 best practices for integrating supportive care practices into the continuum of care for patients with end stage kidney disease (ESKD). In Phase 2 (described in this application), we will conduct a learning collaborative to help up to 15 dialysis and CKD centers implement these best practices. The learning collaborative is based on the IHI Collaborative Model for Achieving Breakthrough Improvement. This model is a tested systematic approach to quality improvement designed to help organizations close the gap between current and future practice based on evidence-based best practices.

The Pathways Project faculty will work with up to 15 change teams at dialysis centers to create a system to identify seriously ill patients with kidney disease; conduct conversations with them so that their values, preferences, and goals for current and future medical treatment are known and respected; assess and address patients' physical, psychological and spiritual needs; and coordinate care throughout the healthcare system so patients receive only the care they want in settings in which they wish to be.

DETAILED DESCRIPTION:
Aim 1: Hold Breakthrough Collaborative for integrating supportive care into kidney care.

To achieve an overall improvement in aligning treatment with patient values and preferences, satisfaction with care, quality of life, and symptom and pain management, Pathways Project Collaborative teams will embark on an 18-month Collaborative beginning spring 2019. Beginning in May 2019, there will be a 4-month observation period to obtain baseline measurements of current supportive care practices at the participating sites. Through the application of the Pathways Project change package, project teams will enhance the delivery of supportive care processes for patients with kidney disease, specifically through the testing and implementation of shared decision-making and advance care planning; systematically identifying seriously ill patients; and providing palliative dialysis to seriously ill patients with advanced Chronic Kidney Disease (CKD) whose goals are not compatible with standard dialysis schedules.

Aim 2: Revise Pathways change package and resources in preparation for dissemination.

In summer 2020, the Pathways Project Advisory Committee, including patient subject matter experts, will revise and strengthen the change package, resources and tools based on the knowledge gained through the Collaborative. The revisions will incorporate the dialysis center/ESCO teams' experience during the collaborative along with the preliminary evaluation results.

Aim 3: Develop strategy for dissemination In fall 2020, the Pathways Project Advisory Committee will develop a strategy to disseminate the revised change package and results of the Collaborative. The dissemination strategy will include outreach to three audiences based on the outcomes of the Pathways Project: 1) the professional and scientific community through presentations at national meetings and articles in peer-reviewed journals; 2) the large dialysis organizations and those who oversee quality of dialysis care including the Forum of ESKD Networks, the individual networks, and the American Health Quality Association; and 3) policy makers including members of Congress and CMS to advocate for changes to improve patient-centered care for patients with kidney disease.

To achieve these aims we will employ three primary tactics:

1. The Institute for Healthcare Improvement (IHI) Breakthrough Collaborative Model - The Collaborative Model is the primary intervention for this project. It has been used to foster successful change adoption in numerous settings with a variety of health problems.
2. The ESCO Model - ESCO stands for ESKD Seamless Care Organizations. ESCO's are a pilot program conducted by CMS to test value-based payment models for dialysis care. The ESCO program brings together economic incentives and organizational innovation factors to create a fertile field for uptake of innovations in patient- and family-centered care in the kidney care continuum. At least four of the participating dialysis centers are part of ESCO demonstration. Three centers (at American Renal Associates) are part of a similar private initiative to provide an integrated care model for ESKD patients.
3. The Pathways Change Package - Provides an evidence-based set of changes and tools collated from the research literature and experiences and efforts of exemplars and organizations that have already successfully adopted supportive care best practices and shown positive outcomes. Justification for the study: Dialysis patients have significant unmet palliative care needs and arguably are the chronic disease patient population who receive the worst end-of-life care because of high intensity care (intensive care unit admission with frequent cardiopulmonary resuscitation, mechanical ventilation and feeding tube use compared to patients with cancer and other chronic diseases) at the end of life with very low referral to hospice. They have a high symptom burden, multiple co-morbid illnesses, and a shortened life expectancy.

Hypothesis: A collaborative quality improvement approach with training of independent dialysis centers and CKD practices in supportive care best practices will lead to improvements in patient and staff-reported outcomes in patient care.

Research Question: Will a collaborative quality improvement approach to spreading supportive care best practices at dialysis centers and affiliated CKD clinics measurably increase the provision of supportive care best practices leading to more effective goal-concordant care?

Relevant background information:

The absence in the United States of a comprehensive medical management without dialysis pathway which is available and selected by about 15% of advanced chronic kidney disease (CKD) patients in other countries is a major deficit in U.S. kidney care. In other ways as well, the current care of patients with advanced CKD in the U.S. is not patient-centered, nor does it utilize supportive care [i] approaches to optimize patients' quality of life. The Pathways Project is seeking to address these deficits through the implementation of a Collaborative.

In a 2013 survey of dialysis center staff, only 4.5% of 487 respondents believed they were presently providing high-quality supportive care including at the end-of-life. When asked what one change could most improve supportive care in their dialysis center, the top choice was "guidelines to help with decision making in seriously ill patients." The second most frequently selected choice was the availability of supportive care consultation to patients. With the exception of a few innovative practices, specialty supportive care consultations are not generally available to patients on dialysis. In those places where supportive care consultation is an option for seriously ill patients on dialysis, nephrologists and their teams typically have not been trained in eliciting shared decision-making, communication, and symptom management skills that would help them deliver primary supportive care.

Shared decision-making is a necessary component to informed consent for patients with advanced CKD. The American Society of Nephrology (ASN) has recommended shared decision-making prior to the initiation of dialysis. Despite ASN's recommendation, shared decision-making-the process in which patients and their family collaborate with healthcare providers to develop a care plan and make decisions about treatments based on patient preferences and values as well as the clinical risks and advantages-is poorly integrated into the care of patients with kidney disease. Most nephrologists express lack of comfort in discussing end-of-life issues. Consequently, most patients with CKD and those on dialysis have little awareness of their prognosis.

Patients older than 75 years are the fastest growing segment of the dialysis population, but these patients, especially if they are frail or have co-morbidities, may not experience a survival benefit from dialysis treatment.The current default is to start elderly patients with advanced kidney disease and multiple co-morbid conditions on dialysis irrespective of their prognosis or likelihood of benefit. The symptom burden for patients with advanced CKD is comparable to that for patients on dialysis, and symptoms are under-recognized and under-treated because of lack of nephrology clinician expertise in supportive care.

The symptom burden of patients on dialysis rivals that of those with cancer, and their five-year survival rate is worse. This tremendous suffering leads to staggering rates of voluntary dialysis withdrawal as high as 35% in the oldest groups, yet hospice and supportive care are underutilized. As a result, patients on dialysis are subjected to more aggressive treatment at the end-of-life than patients with other serious illnesses. Most patients die in the hospital and often after intensive procedures including mechanical ventilation, feeding tube placement, and cardiopulmonary resuscitation. Families of deceased dialysis patients rate the quality of their loved ones' end-of-life care worse than families of those with cancer and other chronic conditions.

There is an urgent need to improve the care of patients with advanced and end stage kidney disease (ESKD). The current situation offers the opportunity to intervene with multiple evidence-based supportive care best practices to transform the care of these seriously ill patients by improving the delivery of supportive care throughout the continuum of kidney disease and making available to seriously ill patients who wish to withdraw from dialysis, delay dialysis, or avoid dialysis, a pathway that offers medical management without dialysis.

[i] In surveys of patients and physicians, they prefer the term supportive care over palliative care. The term palliative care will be used to refer to the specialist title of physicians with board certification in hospice and palliative medicine along with specialist palliative care teams and to the practice of "palliative dialysis" which has a particular definition in the literature. Primary supportive care includes basic communication and symptom management skills provided by other than specialty-trained clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Criteria

  1. Patients at least 18 years old who are currently being treated by participating dialysis center.
  2. Dialysis patients identified as "seriously ill" by screening with "surprise question"- a validated tool that identifies patients with elevated mortality risk. The treating nephrologist or nurse practitioner or dialysis nurse answers whether they would be surprised if the patient died in the next 6 months.

Exclusion Criteria:

1. Patients with impaired cognitive decision making processes as determined by a screening tool.
2. Patients who speak language other than English or Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population of subjects will include dialysis patients who were determined to be seriously ill according to the "surprise question" screening tool. (360 at baseline and 360 at the end of the study 18 months later. This includes about 20 patients for pre-testing the survey.) Facility-level monthly report: One report per dialysis center or CKD practice will be obtained monthly. Reports cover all patients at the site, but data only reported in aggregate.
  Patient level demographic/utilization information. This is collected on all patients who are identified as seriously ill (usually 20% of patients). We expect 300 patients to be identified at baseline (20% of the 1500 total patients).
Sampling Method: Non-Probability Sample
Enrollment: 476 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Patient Reported Quality of Communication | [Time Frame: Baseline (June 2019); Post Intervention- After 3rd Action Period (Late 2020)]
  The primary patient reported outcome for the intervention will be patient reported quality of end of life communication, as measured by the Engelberg quality of communication questionnaire, a subscale on end of life communication.
Change in Comprehensive advance care planning documentation | [Time Frame: Baseline (June 2019); Post Intervention- After 3rd Action Period (Late 2020)]
  The comprehensiveness of advance care planning as documented in dialysis center or CKD clinic chart

SECONDARY OUTCOMES:
Change in Patient reported Outcome Measure: Advance Care Planning Engagement | Baseline (June 2019) and after 3rd Action period (late 2020)
  Additional patient reported outcome measures include the change in advance care planning engagement reported from patient interview from baseline to follow up
Change in Patient Perception of Shared-Decision making | Baseline (June 2019) and after 3rd Action period (late 2020)
  Additional patient reported outcome measures including patient perception of shared-decision making in their kidney health care team, which is reported from the patient interview at baseline and follow-up
Change in patient reported outcome about communication about end-of-life | Baseline (June 2019) and after 3rd Action period (late 2020)
  Additional patient reported outcome measures including communication between patient and health care provider about end of life is included in the patient interview to be used at baseline and follow-up
Change in Dialysis Center or CKD Clinic Staff Perceptions of normalization of the change elements | Before 2nd learning session (September 2019), before 3rd learning session (March 2020) and after 3rd Action Period (Late 2020)
  Staff at each site will complete a validated implementation instrument (NOMAD) measuring normalization of specific elements from the change package.
Change in Dialysis Center or CKD Clinic Staff Perceptions of uptake of change package elements | Before 2nd learning session (September 2019), before 3rd learning session (March 2020) and after 3rd Action Period (Late 2020)
  A second survey measures change in organization-wide staff perception of how well their organization provides supportive care services using a staff survey administered prior to the Collaborative and at the end of the Collaborative. The measurement instrument is a staff survey, the Kidney Supportive Care Implementation Quotient (KSC-IQ), developed by the Pathways team. The KSC-IQ assesses perceived implementation of each change concept in the change package

OTHER OUTCOMES:
Utilization measures: Palliative Dialysis | Measured monthly for 18 months.
  Utilization measures monitored for exploratory purposes include patients using palliative dialysis
Utilization measures: patients withdrawing from dialysis | Measured monthly for 18 months.
  Utilization measures monitored for exploratory purposes include patients patients withdrawing from dialysis
Utilization measures: emergency department visits | Measured monthly for 18 months.
  Utilization measures monitored for exploratory purposes include patients visiting emergency departments
Utilization measures: hospitalizations | Measured monthly for 18 months.
  Utilization measures monitored for exploratory purposes include patients hospitalized
Utilization measures: hospice admissions | Measured monthly for 18 months.
  Utilization measures monitored for exploratory purposes include patients admitted to hospice

CONTACTS AND LOCATIONS:
Overall Officials: Dale E Lupu, PhD, MPH, Principal Investigator — The George Washington University; Alvin Moss, MD, Principal Investigator — West Virginia University
Locations (13):
- United States (13):
  - Kidney Center of Arvada, Arvada, Colorado
  - Thornton Kidney Center, Thornton, Colorado
  - Kidney Center of Westminster, Westminster, Colorado
  - George Washington University, Washington D.C., District of Columbia
  - Washington DC VA Medical Center, Washington D.C., District of Columbia
  - Atlantic Dialysis Astoria, Astoria, New York
  - Rogosin Institute Auburndale, Flushing, New York
  - Atlantic Dialysis Newton, Long Island City, New York
  - Rogosin Institute Manhattan East, New York, New York
  - Atlantic Dialysis Ridgewood, Ridge, New York
  - Rogosin Institute Woodside, Woodside, New York
  - Dallas Nephrology Associates, Dallas, Texas
  - Desoto Regional Dialysis Center, DeSoto, Texas

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Background] Lupu DE, Aldous A, Harbert G, Kurella Tamura M, Holdsworth LM, Nicklas A, Vinson B, Moss AH. Pathways Project: Development of a Multimodal Innovation To Improve Kidney Supportive Care in Dialysis Centers. Kidney360. 2020 Nov 23;2(1):114-128. doi: 10.34067/KID.0005892020. eCollection 2021 Jan 28. PMID 35368811
- [Result] Kurella Tamura M, Holdsworth L, Stedman M, Aldous A, Asch SM, Han J, Harbert G, Lorenz KA, Malcolm E, Nicklas A, Moss AH, Lupu DE. Implementation and Effectiveness of a Learning Collaborative to Improve Palliative Care for Seriously Ill Hemodialysis Patients. Clin J Am Soc Nephrol. 2022 Oct;17(10):1495-1505. doi: 10.2215/CJN.00090122. Epub 2022 Sep 14. PMID 36104084
- [Derived] Holdsworth LM, Stedman M, Gustafsson ES, Han J, Asch SM, Harbert G, Lorenz KA, Lupu DE, Malcolm E, Moss AH, Nicklas A, Kurella Tamura M. "Diving in the deep-end and swimming": a mixed methods study using normalization process theory to evaluate a learning collaborative approach for the implementation of palliative care practices in hemodialysis centers. BMC Health Serv Res. 2023 Dec 11;23(1):1384. doi: 10.1186/s12913-023-10360-7. PMID 38082293
- [Derived] Moss AH, Harbert G, Aldous A, Anderson E, Nicklas A, Lupu DE. Pathways Project Pragmatic Lessons Learned: Integrating Supportive Care Best Practices into Real-World Kidney Care. Kidney360. 2023 Dec 1;4(12):1738-1751. doi: 10.34067/KID.0000000000000277. Epub 2023 Oct 27. PMID 37889550
- See also: Pathways Project Website — https://www.nursing.gwu.edu/pathways-project

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/37/NCT04125537/Prot_SAP_000.pdf